CLINICAL TRIAL: NCT03651583
Title: Pilot Study Examining the Efficacy of Kiko Exercises on the Prevention of Migraine Headaches
Brief Title: Examining the Efficacy of Kiko Exercises on the Prevention of Migraine Headaches
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Regional Clinical Research (Other)
Responsible Party: Principal Investigator, Victor Elinoff MD, Principal Investegator, Regional Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Kiko Protocol 01
Record Dates: First submitted 2014-11-05; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Migraine Headache
Keywords: Migraine; Kiko; Qigong; Relaxation; Exercise
MeSH Terms: conditions — Migraine Disorders; Motor Activity | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot Trial (Other): Behavioral Intervention Kiko exercises-combines breathing and movement all study subjects no placebo or control group
  Interventions: Behavioral: Kiko exercises-combines breathing and movement

INTERVENTIONS:
Behavioral: Kiko exercises-combines breathing and movement

SUMMARY:
This pilot study hopes to show that after 3 months of Kiko training, Kiko naive patients with migraine will have a decrease in the frequency and severity of their migraines.

DETAILED DESCRIPTION:
3.1 Study Design

Eligible subjects in this pilot study will be taught a series of Kiko exercises. Subjects who meet inclusion and exclusion criteria at the screening visit will be given a diary in which they will document their migraine frequency and severity for one month. Once subject diaries are complete, subjects will meet for a group lesson to learn the background of Kiko and study exercises. A DVD or videotape will be issued for subjects to use during practice at home. Subjects will maintain a diary of their migraine headaches, as well as a diary of their exercise routines. Subjects will meet weekly to reinforce training and encourage training continuation. Diaries will be collected at the end of the first, second, and third months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 70 years of age, with at least a 1-year history of migraine headaches
* With or without aura, (IHS criteria 1.1 and 1.2), who have experienced at least 4 migraines a month, or 2-3 migraines a month that last 2-3 days per attack in each of the 3 months prior to screening.
* The subjects must be naïve to Kiko and Qigong training.

Exclusion Criteria:

1. Subject has any cardiac condition, as determined by the investigator, that would preclude safe participation in a low level exercise program.
2. Uncontrolled hypertension at screening (sitting systolic pressure >160 mmHg, diastolic pressure >95 mmHg.)
3. Subject has had tension-type headaches, >15 days/month in any of the 3 months prior to screening.
4. Subject has more than 8 migraines per month, or more than 16 days of migraine per month.
5. Subject is pregnant or expects to become pregnant during the course of the trial.
6. Subject has substance or alcohol abuse within the the last year which, in the investigator's judgement, will interfere with the study conduct, cooperation or evaluation and interpretation of the study results.
7. Subject has any concurrent medical or psychological condition that, in the investigator's opinion, may affect the interpretation of efficacy or safety data or which otherwise contraindicates participation in the trial.
8. Subject has participated in an investigational drug trial within the previous 4 weeks.
9. Subject uses pain medication in excess of 40 doses of over the counter medication and/or prescription pain medication per month to treat headaches of any type.
10. Subject is unable to differentiate between migraine and non-migraine headaches.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change in Migraine Frequency and Severity from Baseline | 3 months
  Change in Migraine Frequency and Severity from Baseline on LIkert Scale 1-4

SECONDARY OUTCOMES:
Change in number of headache free days | 3 months
  Change in number of headache free days from baseline based on Diary Data
Change in number of migraine free days | 3 months
  Change in number of Migraine free days from baseline based on diary data
Change in overall quality of life | 3 month
  Change in quality of life from baseline based on LIkert scale 1-2
Subject satisfaction with Kiko training | 3 months
  Satisfaction measurement of training based on LIkert scale 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Victor Elinoff, MD, Principal Investigator — Regional Clinical Research
Locations (1):
- Endwell Family Physicians, Endwell, New York, United States